CLINICAL TRIAL: NCT06946147
Title: Assessment of Temporomandibular Joint Function Across Different Trimesters of Pregnancy
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Zaghloul Mohammed, Principal investigator, Cairo University
Other Study IDs: P.T.REC/012/005674
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Temporomandibular; Functional Disturbance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women: Assessment of Temporomandibular Joint Function will be conducted in pregnant women through different trimesters of pregnancy at specific measuring times:
  Baseline: early first trimester (before 12 weeks of gestation). Second trimester: between 18 and 21 weeks of gestation. Third trimester: between 31 and 34 weeks of gestation.
- Non- pregnant women: Assessment of Temporomandibular Joint Function will be conducted in non-pregnant healthy women.

INTERVENTIONS:
Other:

SUMMARY:
This study will be conducted to assess Temporomandibular Joint (TMJ) function across different trimesters of pregnancy.

DETAILED DESCRIPTION:
Pregnancy is a physiological state that can potentially influence the function and biomechanics of the Temporomandibular Joint (TMJ) due to hormonal changes, weight gain, and other associated factors. TMJ disorders are a common problem affecting a significant proportion of the population, with potential impacts on chewing, speaking, and other daily functions, significantly affecting a pregnant woman's quality of life.

Limited research has been conducted to comprehensively evaluate the changes in TMJ function and proprioception (repositioning accuracy) across different trimesters of pregnancy. By identifying and understanding the specific impacts of different trimesters of pregnancy on TMJ function, this study aims to provide insights that can help in the early detection and effective management of TMJ disorders. This, in turn, can improve the overall well-being and comfort of pregnant women, contributing to a more positive pregnancy experience.

Moreover, physiotherapists currently have limited guidelines specifically tailored for managing TMJ dysfunction in pregnant patients. This study aims to fill this gap by providing evidence-based insights into the mechanisms and risk factors associated with TMJ dysfunction during pregnancy. The findings can inform the development of clinical guidelines and therapeutic protocols that address the unique needs of pregnant women, ensuring safer and more effective care.

ELIGIBILITY:
Inclusion Criteria:

All women will be pregnant with a single baby. Their ages will range from 20 to 35 years old. Their parity will range from 1 to 2. Their body mass index will range from 20 to 30kg2.

Exclusion Criteria:

All women will not suffer from any TMJ disorder or orofacial pain before pregnancy.

All women will not suffer from any severe dental pathology. All women will not suffer from high-risk pregnancy (hyperemesis gravidarum, gestational diabetes).

All women will not suffer from any systemic illnesses.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Twenty pregnant women and twenty non-pregnant women will participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Mouth Opening (Eyes Open) | 5 months
  The woman opens her mouth maximally. The vertical distance between the upper and lower central incisors is measured using a caliper. One-third of the full temporomandibular joint range of motion (ROM) is used as functional ROM. The caliper is adjusted to this range. The woman practices the motion three times, then performs it actively three times with eyes open. Mean absolute joint position error (JPE) is recorded.
Mouth Opening (Eyes Closed) | 5 months
  The woman opens her mouth maximally. The vertical distance between the upper and lower central incisors is measured using a caliper. One-third of the full temporomandibular joint range of motion (ROM) is used as functional ROM. The caliper is adjusted to this range. The woman practices the motion three times, then performs it actively three times with eyes closed. Mean absolute joint position error (JPE) is recorded.
Right Lateral Movement (Eyes Open): | 5 months
  From rest, the woman moves her jaw to the right. The horizontal distance between upper and lower incisors is measured. Functional range of motion ROM is calculated (one-third of full ROM). She practices then actively performs the movement three times. Joint position error (JPE) is recorded.
Right Lateral Movement (Eyes Closed) | 5 months
  From rest, the woman moves her jaw to the right. The horizontal distance between upper and lower incisors is measured. Functional range of motion (ROM) is calculated (one-third of full ROM). She practices then actively performs the movement three times but with eyes closed. Joint position error (JPE) is recorded.
Left Lateral Movement (Eyes Open) | 5 months
  From rest, the woman moves her jaw to the left. The horizontal distance between upper and lower incisors is measured. Functional range of motion (ROM) is calculated (one-third of full ROM). She practices then actively performs the movement three times.Joint position error (JPE) is recorded.
Left Lateral Movement (Eyes Closed) | 5 months
  rom rest, the woman moves her jaw to the left. The horizontal distance between upper and lower incisors is measured. Functional range of motion (ROM) is calculated (one-third of full ROM). She practices then actively performs the movement three times but with eye closed. Error of JPE is recorded.
Jaw protrusion (Eyes Open) | 5 months
  From rest, the woman moves her jaw forward. Distance between upper and lower incisors is measured. Functional range of motion (ROM) is calculated. Movement is practiced and repeated three times. Joint position error (JPE) is recorded.
Jaw protrusion (Eyes Closed) | 5 months
  From rest, the woman moves her jaw forward. Distance between upper and lower incisors is measured. Functional range of motion (ROM) is calculated. Movement is practiced and repeated three times but with closed eyes. Joint position error (JPE) is recorded.

SECONDARY OUTCOMES:
Assessment of severity of temporomandibular joint dysfunction | 5 months
  The Fonseca's questionnaire follows the characteristics of a multidimensional evaluation. It is composed of 10 questions, which include checking for the presence of pain in the TMJ, head, back, and while chewing, parafunctional habits, movement limitations, joint clicking, perception of malocclusion, and sensation of emotional stress. The volunteers will be informed that the 10 questions should be answered with "yes," "no," and "sometimes," and that only one answer should be marked for each question. Each answer choice is assigned a score (typically 10 for "yes," 5 for "sometimes," and 0 for "no"). The total score is then calculated by summing the scores for all questions. Higher scores indicate a greater likelihood of TMJ dysfunction
Assessment of temporomandibular joint pain | 5 months
  The level of pain in the temporomandibular joint will be assessed through the visual analogue scale (VAS). The VAS is a pain rating scale, whose scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and "worst pain" on the right end of the scale (10 cm). Measurements from the starting point (left end) of the scale to the participants' marks will be recorded in centimeters and will be interpreted as their pain level.

CONTACTS AND LOCATIONS:
Overall Officials: HAZEM EL ASHMAWY, Professor, Study Director — Cairo University; Doaa Osman, Professor, Study Chair — Cairo University
Locations (1):
- Maha Zaghloul mohammed, Cairo, Egypt